CLINICAL TRIAL: NCT05502172
Title: Evaluation of the Effectiveness of Nutritional Intervention With Fish-derived Lipids in Improving Antiviral Immunity in Healthy People
Brief Title: Effects of Nutritional Intervention With Fish-derived Lipids in Improving Antiviral Immunity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marinex International Sp. z o.o. (Industry)
Responsible Party: Principal Investigator, Natalia Lewkowicz, Professor, Medical University of Lodz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RNN/52/22/KE
Record Dates: First submitted 2022-08-04; First posted 2022-08-16 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Nutrition, Healthy
Keywords: fish oil; antiviral immune reponse
MeSH Terms: interventions — Fish Oils

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- fish oil (Experimental): Healthy individuals will be taking the composition of fish-derived oils BioMarine®Medical Immuno & Neuro Lipids at a dose of 0.5 ml / kg body weight per day in two / three divided doses for 90 days.
  Interventions: Dietary Supplement: fish oil

INTERVENTIONS:
Dietary Supplement: fish oil — healthy individuals will be taking the composition of fish-deraivd oils BioMarine®Medical Immuno & Neuro Lipids at a dose of 0.5 ml / kg body weight per day in two / three divided doses for 90 days.
  Other Names: BioMarine®Medical Immuno&Neuro Lipids

SUMMARY:
The aim of the study is to evaluate the effects of fish-derived lipids on antiviral immunity in healthy individuals. The study will be conducted on a group of 30 healthy volunteers recruited at the Department of Periodontology and Oral Diseases of the Medical University of Lodz. These people will take a composition of fish-derived oils (BioMarine®Medical Immuno & Neuro Lipids) at a dose of 0.5 ml / kg body weight per day in two / three divided doses for 90 days. BioMarine®Medical Immuno & Neuro Lipids is food for special medical purposes. At baseline and after 90 days, blood samples will be taken from the test subjects in order to evaluate the selected parameters of antiviral immunity.

DETAILED DESCRIPTION:
The proposed clinical trial involving a nutritional intervention aims to assess the effect of a composition of fish oils containing, inter alia, WWKT omega-3 EPA and DHA, alkylglycerols and squalene on selected parameters of antiviral immunity in healthy people. The proposed daily dose of BioMarine®Medical Immuno & Neuro Lipids is 0.5 ml / kg b.w., which in practice for a person weighing 60 kg will mean a daily consumption of 30 mL of oil (including 1.6 g EPA, 9.1 g DHA, 2 5 g of alkylglycerols and 2.6 g of squalene).

At baseline, 15 ml of blood will be drawn in order to determine the parameters of the antiviral response.

The following immunological parameters will be tested:

1. NK cell activity using a mixed culture of PBMC with target cells (ability to inhibit tumor cell proliferation) assessed by flow cytometry.
2. Absolute number and percentage of NK cells (CD16 + CD56 +), cytotoxic (CD8 +), helper (CD4 +) lymphocytes, B (CD19 +) lymphocytes in the total pool of peripheral blood mononuclear cells (PBMC) by flow cytometry.
3. Ability of isolated PBMCs to synthesize INF-α, INF-β, INF-γ, IL-6 and TNF without and after polyclonal stimulation (PHA) and SARS-CoV-2 proteins (nucleocapside protein, SARS-CoV-2 spike protein ) in 42 h culture based on the determination of the level of protein released into the culture fluid and on the basis of mRNA expression for these factors. Analysis of PBMC post-culture supernatants (CBA technique with flow cytometer and gene expression analysis by qPCR).
4. Analysis of the composition of serum lipids and in PBMC lyophilisates after culture.

Blood sampling will be repeated after 90 days in order to determine the influence of the fish oils on the tested parameters.

ELIGIBILITY:
Inclusion Criteria:

* absence of systemic diseases;
* no medications taken on a regular basis;
* correct body weight in relation to height - 18.5 ≤ BMI ≤ 24.9

Exclusion Criteria:

* lack of consent the patient'sto the examination.
* pregnant and lactating women;
* smokers or non-smokers for less than 5 years;
* any vaccinations in the period shorter than 1 month before the start of the study or planned during the study;
* lack of declaration on reducing fats in the diet and avoiding highly processed fats and fried products.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2022-11-18 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-07-12 (Actual)

PRIMARY OUTCOMES:
Change in peripheral blood NK cell activity | baseline, 90 days
  NK cell activity using a mixed culture of PBMC with target cells (ability to inhibit tumor cell proliferation) assessed by flow cytometry.
Change in the number and percentage of peripheral blood NK cells, CD8 cells, CD4 cells, CD19 cells | baseline, 90 days
  Absolute number and percentage of NK cells (CD16 + CD56 +), cytotoxic (CD8 +), helper (CD4 +) lymphocytes, B (CD19 +) in the total pool of peripheral blood mononuclear cells (PBMC) by flow cytometry.
Change in the production of cytokines (INF-α, INF-β, INF-γ, IL-6 and TNF) by peripheral blood mononuclear cells | baseline, 90 days
  Ability of isolated PBMCs to synthesize INF-α, INF-β, INF-γ, IL-6 and TNF without and after polyclonal stimulation (PHA) and SARS-CoV-2 proteins (nucleocapside protein, SARS-CoV-2 spike protein ) in 42 h culture based on the determination of the level of protein released into the culture fluid and on the basis of mRNA expression for these factors. Analysis of PBMC post-culture supernatants (CBA technique with flow cytometer and gene expression analysis by qPCR).

SECONDARY OUTCOMES:
Change in serum lipid content | baseline, 90 days
  Analysis of lipid composition using gas/spectrum chromotography
Change in in lipid content in PBMC lyophilisates | baseline, 90 days
  Analysis of lipid composition using gas/spectrum chromotography

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Lewkowicz, prof., Principal Investigator — Medical University of Lodz
Locations (1):
- Department of Periodontology and Oral Diseases, Lodz, Poland

IPD SHARING:
Plan to Share IPD: No